CLINICAL TRIAL: NCT02668562
Title: Reassessment of Anti-Platelet Therapy Using InDividualized Strategies -Ticagrelor in Patients With Acute Coronary Syndromes Treated by Coronary Artery Bypass Graft Surgery - A Pharmacodynamic and Clinical Study to Decrease Bleeding Risks and Ischemic Complications - The RAPID-TITRATE CABG Study
Brief Title: Timing of Coronary Artery Bypass Surgery Among Patients With Acute Coronary Syndromes Initially on Ticagrelor
Acronym: RAPID CABG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20150656
Record Dates: First submitted 2016-01-06; First posted 2016-01-29 (Estimated); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Acute Coronary Syndrome
Keywords: acute coronary syndrome; coronary artery bypass surgery; ticagrelor; antiplatelet therapy; platelet function testing
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early CABG (Experimental): Patients to undergo early CABG
  Interventions: Procedure: Early CABG (Day 2-3 after ticagrelor discontinuation)
- Delayed CABG (Active Comparator): Patients to undergo delayed CABG
  Interventions: Procedure: Delayed CABG (Day 5-7 after ticagrelor discontinuation)

INTERVENTIONS:
Procedure: Early CABG (Day 2-3 after ticagrelor discontinuation) — Timing for CABG after ticagrelor discontinuation
  Arms: Early CABG
Procedure: Delayed CABG (Day 5-7 after ticagrelor discontinuation) — Timing for CABG after ticagrelor discontinuation
  Arms: Delayed CABG

SUMMARY:
Ticagrelor, a more potent P2Y12 inhibitor, has been shown to reduce major adverse cardiac events (MACE) in acute coronary syndromes (ACS). It is increasingly used as a first line therapy in ACS. However, more potent P2Y12 inhibition has been associated with increased bleeding. This may be of particular concern for patients with ACS who require coronary artery bypass surgery (CABG). In particular, the timing for cessation of ticagrelor before proceeding to CABG is unclear. RAPID TITRATE CABG is a randomized vanguard study to evaluate the feasibility and preliminary safety of a strategy of early versus delayed CABG in ACS patients initially treated with ticagrelor and to identify potential mechanisms underlying benefits or complications of early bypass surgery.

ELIGIBILITY:
Inclusion Criteria:

* ACS patient referred for CABG and have received >= 1 dose of ticagrelor before decision for CABG made

Exclusion Criteria:

Patients are excluded if they:

* refuse consent for enrollment
* are deemed to require immediate CABG (Day 0 or day 1)
* have a ST-elevation myocardial infarction (STEMI )initially treated with primary PCI
* are undergoing concurrent valve surgery
* are intolerant or allergic to aspirin
* have been on an oral anticoagulant (including a vitamin K antagonist or a NOAC)
* received adjuvant therapy with a glycoprotein IIbIIIa inhibitor
* have a co-morbidity with life-expectancy of < 1 year
* have active bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2021-04-09 (Actual); Study Completion 2022-03-09 (Actual)

PRIMARY OUTCOMES:
Severe-massive bleeding | 24 hours post CABG
  Class 3 or 4 UDPB (universal definition for peri-operative bleeding)
12-hour chest tube drainage | 12 hours post CABG
  Chest tube drainage in the first 12 hours after bypass surgery

SECONDARY OUTCOMES:
Other major bleeding criteria (BARC) | 48 hours post CABG
  Bleeding Academic Research Consortium (BARC) CABG-related (Type 4) bleeding
Other major bleeding criteria (TIMI) | 48 hours post CABG
  TIMI major/minor CABG bleeding
Other major bleeding criteria (CABG related life threatening bleed) | 48 hours post CABG
  CABG-related life-threatening bleed including: cardiac tamponade, all intracranial bleeding
Transfusion (RBC) | 48 hours post CABG
  Red Blood Cell (RBC) transfusion (in Units)
Transfusion (Platelet) | 48 hours post CABG
  Platelet transfusion (in Units)
Peri-operative biomarker rise | 48 hours post CABG
  CK, troponin rise post CABG
Number of Patients with Major Adverse Cardiovascular Events (MACE) (To be collected but blinded to investigators,as this data will be carried from the vanguard study into a future definitive clinical trial). | 6 months and 1 year
  MACE defined as composite of cardiovascular death, recurrent myocardial infarction, stroke, refractory ischemia, or urgent unplanned revascularization
Number of Patients with Individual Components of Major Adverse Cardiovascular Events (MACE) (To be collected but blinded to investigators,as this data will be carried from the vanguard study into a future definitive clinical trial). | 6 months and 1 year
  cardiovascular death, recurrent myocardial infarction, stroke, refractory ischemia, or urgent unplanned revascularization
P2Y12 Reactivity Units (PRU) as a continuous variable | Baseline (at CABG), 24, 48, 72 hours post CABG
  Platelet Function as Measured by VerifyNow P2Y12 assay
ADP-induced Aggregation (AU) as a continuous variable | Baseline (at CABG), 24, 48, 72 hours post CABG
  Platelet Function as Measured by Multiplate analyzer

CONTACTS AND LOCATIONS:
Overall Officials: Derek So, MD FRCPC FACC, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (2):
- Canada (2):
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Montreal Heart Institute, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] So DYF, Wells GA, Lordkipanidze M, Chong AY, Ruel M, Perrault LP, Le May MR, Sun L, Tran D, Labinaz M, Glover C, Russo J, Welman M, Chan V, Chen L, Bernick J, Rubens F, Tanguay JF; RAPID CABG Investigators. Early vs Delayed Bypass Surgery in Patients With Acute Coronary Syndrome Receiving Ticagrelor: The RAPID CABG Randomized Open-Label Noninferiority Trial. JAMA Surg. 2025 Apr 1;160(4):387-394. doi: 10.1001/jamasurg.2024.7066. PMID 39969871